CLINICAL TRIAL: NCT02575768
Title: Reduced Myocardial Flow Reserve in Exertional Angina With Severe Aortic Stenosis and Normal Coronary Arteries: Insight From Prospective Observational Adenosine-stress Cardiac Magnetic Resonance Imaging Study
Brief Title: Myocardial Flow Reserve in Severe AS Without Obstructive Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-01-014
Record Dates: First submitted 2015-08-31; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2012-06

CONDITIONS: Chest Pain; Severe Aortic Stenosis
MeSH Terms: conditions — Chest Pain; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Severe AS: asymptomatic: Asymptomatic
  Interventions: Other: Adenosine-stress cardiac magnetic resonance imaging
- Severe AS: pure angina: Presence of exertional chest pain
  Interventions: Other: Adenosine-stress cardiac magnetic resonance imaging
- Normal controls: Healthy controls
  Interventions: Other: Adenosine-stress cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Adenosine-stress cardiac magnetic resonance imaging — undergoing adenosine-stress cardiac magnetic resonance imaging

SUMMARY:
Exertional angina is common symptom in patients with severe aortic stenosis (AS) without obstructive coronary artery disease (CAD). Although reduced myocardial flow reserve is one of the proposed explanations for angina, little is known about the pathophysiology.

This study aimed that adenosine-stress cardiac magnetic resonance can be used for the assessment of myocardial perfusion reserve and suggest the pathophysiology of development of angina in patients with severe AS without obstructive CAD.

ELIGIBILITY:
Inclusion Criteria:

1. severe AS
2. normal LV ejection fraction (EF ≥ 50%)

Exclusion Criteria:

1. age <18
2. LVEF < 50% in echocardiography
3. concomitant other valvular disease of moderate or severe severity
4. previous aortic valve replacement
5. symptomatic patients other than chest pain
6. obstructive CAD (>30% luminal stenosis in at least one coronary artery on coronary angiography)
7. history of myocardial infarction or acute coronary syndrome
8. contraindication to adenosine
9. any absolute contraindication to CMR
10. estimated glomerular filtration rate <30 mL/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who had severe AS and normal LV ejection fraction (EF ≥ 50%) in transthoracic echocardiography were included in the investigators' prospective study. Severe AS was defined as aortic valve area index less than 0.6 cm2/m2 as previously published.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Values of the myocardial perfusion reserve index (MPRI) | Day 1
  Signal intensity-time curves were generated for all segments and the maximum upslope of the LV myocardium divided by the maximum upslope of the LV cavity. MPRI [upslopestress(corrected)/upsloperest(corrected)] was calculated dividing the segmental upslope value during adenosine and rest. Whole (average of all myocardial segments) MPRI were calculated.

REFERENCES:
- [Background] American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; Bonow RO, Carabello BA, Kanu C, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B. ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (writing committee to revise the 1998 Guidelines for the Management of Patients With Valvular Heart Disease): developed in collaboration with the Society of Cardiovascular Anesthesiologists: endorsed by the Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. Circulation. 2006 Aug 1;114(5):e84-231. doi: 10.1161/CIRCULATIONAHA.106.176857. No abstract available. PMID 16880336
- [Background] Silaruks S, Clark D, Thinkhamrop B, Sia B, Buxton B, Tonkin A. Angina pectoris and coronary artery disease in severe isolated valvular aortic stenosis. Heart Lung Circ. 2001;10(1):14-23. doi: 10.1046/j.1444-2892.2001.00060.x. PMID 16352020
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):e57-185. doi: 10.1016/j.jacc.2014.02.536. Epub 2014 Mar 3. No abstract available. PMID 24603191
- [Derived] Ahn JH, Kim SM, Park SJ, Jeong DS, Woo MA, Jung SH, Lee SC, Park SW, Choe YH, Park PW, Oh JK. Coronary Microvascular Dysfunction as a Mechanism of Angina in Severe AS: Prospective Adenosine-Stress CMR Study. J Am Coll Cardiol. 2016 Mar 29;67(12):1412-1422. doi: 10.1016/j.jacc.2016.01.013. PMID 27012401